CLINICAL TRIAL: NCT03291652
Title: Morphology of Advanced Symptomatic Cerebral Plaques With High Embolic Potential
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Leung Wai Hong Thomas, Professor, Chinese University of Hong Kong
Other Study IDs: crec no. 2011.021
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Stroke; Atheroscleroses, Cerebral
Keywords: Ischemic Stroke; atherosclerosis; Plaque morphology; DSA/3DRA
MeSH Terms: conditions — Ischemic Stroke; Intracranial Arteriosclerosis; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic stroke patient: DSA and 3DRA will be performed with access through a 4F sheath at the right femoral artery. Angiograms of intracranial arteries will be obtained by contrast injection at internal carotid artery and vertebral artery ostium from a 4F H1 catheter. Each injection will contain 10ml of iopaminro 300 diluted in 1:1 with normal saline. Each angiographic run will capture a complete series of images from the arterial phase to the end of the venous phase. A 3-dimensional rotational angiogram (a scan time of 4 seconds with 120 images) will be obtained for evaluation of plaque morphology.
  2. The access site will be closely observed for hemostasis after the procedure. The neurological status and renal function will be monitored.
  Diagnosis procedure: DSA/3DRA
  Interventions: Diagnostic Test: DSA/3DRA
- Asymptomatic stroke patient: DSA and 3DRA will be performed with access through a 4F sheath at the right femoral artery. Angiograms of intracranial arteries will be obtained by contrast injection at internal carotid artery and vertebral artery ostium from a 4F H1 catheter. Each injection will contain 10ml of iopaminro 300 diluted in 1:1 with normal saline. Each angiographic run will capture a complete series of images from the arterial phase to the end of the venous phase. A 3-dimensional rotational angiogram (a scan time of 4 seconds with 120 images) will be obtained for evaluation of plaque morphology.
  2. The access site will be closely observed for hemostasis after the procedure. The neurological status and renal function will be monitored.
  Diagnosis procedure: DSA/3DRA
  Interventions: Diagnostic Test: DSA/3DRA

INTERVENTIONS:
Diagnostic Test: DSA/3DRA — DSA/3DRA

SUMMARY:
The study is to attain early recognition of the unstable plaques which have an imminent embolic risk in patients with intracranial atherosclerotic disease (IAD).

DETAILED DESCRIPTION:
Potential candidates will undergo a cranial MRI and MR angiography. Patients who are found signal void in a relevant intracranial internal carotid artery or middle cerebral artery will proceed to a 30-minute TCD monitoring for MES an angiograms will be analyzed by investigators blind to subjects' clinical information. All recruited patients will receive standard medical therapy throughout the investigation period.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for the Symptomatic Group:

  1. Patient is 30 to 85 years of age, inclusive.
  2. Patients who have an acute infarct in diffusion-weighted MRI compatible with artery-to-artery thrombo-embolism, a relevant intracranial atherosclerotic stenosis ≥60%, and MES detected by TCD.
  3. Patient who has no contra-indication for the proposed imaging tests.
  4. Patient understands the purpose and requirements of the study, and has provided an informed consent.
* Inclusion Criteria for the Asymptomatic Group:

  1. Patient is 30 to 85 years of age, inclusive.
  2. Patient who has a high-grade (>60%) intracranial stenosis (signal void in MR angiography) but without infarct in the corresponding vascular territory in DWI or T2-weighted sequence.
  3. Patient has no MES detected on TCD examination.
  4. Patient who has no contra-indication for the proposed imaging tests.
  5. Patient understands the purpose and requirements of the study, and has provided an informed consent.

Exclusion Criteria:

Subject who meets one or more of the following criteria cannot be recruited in the study:

1. Stroke etiology uncertain or unrelated to intracranial atherosclerosis, such as cardioembolism, Moyamoya disease, small vessel disease, etc.
2. A tandem stenosis >50% at proximal internal carotid artery.
3. Bleeding propensity: active peptic ulcer disease, major systemic hemorrhage within 30 days, thrombocytopenia (platelets <100 x 109/L), coagulopathy (INR >1.5).
4. A medical condition that would not allow the patient to adhere to the protocol or complete the study.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who admitted to Prince of Wales Hospital for acute stroke will be screened for eligibility.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2010-02 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The plaque morphology of high-risk IAD may be distinct from the silent ones. | Dec, 2020
  The morphological attributes (surface outline, angulations and plaque volume) and collateral grading will be compared between symptomatic and asymptomatic group.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wai Hong LEUNG, FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No